CLINICAL TRIAL: NCT03141801
Title: Blood Flow Restriction Training to Improve Muscle Strength and Function Following Anterior Cruciate Ligament Injury
Brief Title: Blood Flow Restriction to Improve Muscle Strength After ACL Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00110455
Record Dates: First submitted 2017-04-17; First posted 2017-05-05 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL; Knee; Muscle
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eccentric Exercise with Delfi Blood Flow Restriction Training (Experimental): Patients randomized to the eccentric exercise + blood flow restriction training group will receive eccentric exercise two times per week for 8 weeks, beginning 8-12 weeks after anterior cruciate ligament reconstruction. Patients will completed the exercise with knee range of motion limited to 20-60 degrees of knee flexion and will train at an intensity equal to 70% of their eccentric 1-repetition maximum for 4 sets of 10 repetitions. During exercise, patients will have the DELFI personalized tourniquet system applied over the quadriceps to restrict blood flow. The tourniquet will be set to a limb occlusion pressure of 80%.
  Interventions: Device: DELFI PTS Personalized Tourniquet System for Blood Flow Restriction Training; Other: Eccentric Exercise with BLAST Leg Press System
- Concentric Exercise with Delfi Blood Flow Restriction Training (Experimental): Patients randomized to the concentric exercise group will receive concentric exercise two times per week for 8 weeks, beginning 8-12 weeks after anterior cruciate ligament reconstruction. Patients will completed the exercise with knee range of motion limited to 20-60 degrees of knee flexion and will train at an intensity equal to 70% of their concentric 1-repetition maximum for 4 sets of 10 repetitions.
  Interventions: Device: DELFI PTS Personalized Tourniquet System for Blood Flow Restriction Training; Other: Concentric Exercise with BLAST Leg Press System
- Eccentric Exercise (Active Comparator): Patients randomized to the eccentric exercise group will receive eccentric exercise two times per week for 8 weeks, beginning 8-12 weeks after anterior cruciate ligament reconstruction. Patients will completed the exercise with knee range of motion limited to 20-60 degrees of knee flexion and will train at an intensity equal to 70% of their eccentric 1-repetition maximum for 4 sets of 10 repetitions.
  Interventions: Other: Eccentric Exercise with BLAST Leg Press System
- Concentric Exercise (Active Comparator): Patients randomized to the concentric exercise group will receive concentric exercise two times per week for 8 weeks, beginning 8-12 weeks after anterior cruciate ligament reconstruction. Patients will completed the exercise with knee range of motion limited to 20-60 degrees of knee flexion and will train at an intensity equal to 70% of their concentric 1-repetition maximum for 4 sets of 10 repetitions. During exercise, patients will have the DELFI personalized tourniquet system applied over the quadriceps to restrict blood flow. The tourniquet will be set to a limb occlusion pressure of 80%.
  Interventions: Other: Concentric Exercise with BLAST Leg Press System

INTERVENTIONS:
Device: DELFI PTS Personalized Tourniquet System for Blood Flow Restriction Training — cuff is inflated to 80% of an individuals limb occlusion pressure
  Other Names: Kaatsu Training
  Arms: Concentric Exercise with Delfi Blood Flow Restriction Training; Eccentric Exercise with Delfi Blood Flow Restriction Training
Other: Eccentric Exercise with BLAST Leg Press System — 4 sets of 10 repetitions of an eccentric leg press exercise performed at 70% of the 1 repetition maximum
  Arms: Eccentric Exercise; Eccentric Exercise with Delfi Blood Flow Restriction Training
Other: Concentric Exercise with BLAST Leg Press System — 4 sets of 10 repetitions of an concentric leg press exercise performed at 70% of the 1 repetition maximum
  Arms: Concentric Exercise; Concentric Exercise with Delfi Blood Flow Restriction Training

SUMMARY:
Quadriceps muscle weakness is a common consequence following anterior cruciate ligament (ACL) injury and reconstruction. Maximizing quadriceps strength following ACL injury is significant as diminished quadriceps strength has been linked to the osteoarthritis that affects over 50% of surgically reconstructed limbs. Given that knee joint health following ACL injury is predicated on restoring quadriceps strength, identifying treatment approaches capable of improving strength is paramount. Blood flow restriction training (BFRT) is a method where oxygen to the muscle is intentionally reduced during exercise/rehabilitation and may lead to more timely and substantial strength gains. In the proposed project, we will examine the efficacy of BFRT in patients who have undergone ACL reconstruction and suffer from substantial quadriceps weakness.

DETAILED DESCRIPTION:
Quadriceps muscle weakness is a common consequence following anterior cruciate ligament (ACL) injury and reconstruction. Maximizing quadriceps strength following ACL injury is significant as diminished quadriceps strength has been linked to the osteoarthritis that affects over 50% of surgically reconstructed limbs. Given that knee joint health following ACL injury is predicated on restoring quadriceps strength, identifying treatment approaches capable of improving strength is paramount. Blood flow restriction training (BFRT) is a method whereby oxygen to the muscle is intentionally reduced during exercise/rehabilitation and may lead to more timely and substantial strength gains. In the proposed project, we will examine the efficacy of BFRT in patients who have undergone ACL reconstruction and suffer from quadriceps weakness. This project will have a randomized clinical trial design. Sixty patients that have torn their ACL and plan to undergo surgical reconstruction will be randomized into one of four groups: 1) eccentric exercise; 2) concentric exercise; 3) eccentric exercise with blood flow restriction; or 4) concentric exercise with blood flow restriction. All patients regardless of randomization assignment will also receive standard of care ACL rehabilitation. Approximately 6 weeks after ACL reconstruction surgery, patients will begin to receive the study interventions which will last for 8 weeks. The concentric exercise will be a leg press exercise done on a conventional leg press machine, while the eccentric exercise will be a leg press exercise done on a device designed to elicit eccentric muscle contractions. Patients will train at 70% of their 1 repetition maximum and will complete 4 sets of 10 contractions at each session (2 sessions/week). For patients randomized to the BFRT groups they will complete the leg press exercise while blood flow the the quadriceps muscle is restricted with a BFRT device (Delfi Personalized Tourniquet System for Blood Flow Restriction). We will quantify our dependent variables prior to surgical reconstruction, 6 weeks post-operatively (before study intervention starts), 14 weeks post-operatively (immediately after study intervention ends), and time of physician discharge from rehabilitation (e.g. time medical clearance for return to activity). The primary outcome is isokinetic quadriceps strength. We hypothesize that patients who complete eccentric exercise along with blood flow restriction training will realize the greatest gains in muscle strength.

The DELFI PTS Personalized Tourniquet system is exempt from premarket notification and is therefore not subject to 510(k)

ELIGIBILITY:
Inclusion Criteria:

1. suffered an acute, complete ACL rupture as confirmed by MRI
2. scheduled to undergo ACL reconstruction
3. scheduled to undergo ACL reconstruction with a surgeon affiliated with MedSport (University of Michigan Orthopaedic Clinic)
4. willing to undergo rehabilitation through MedSport (University of Michigan Orthopaedic Clinic) 5)) Willingness to participate in testing and follow-up as outlined in the protocol

6) English-speaking

Exclusion Criteria:

1. inability to provide written informed consent (or assent)
2. female subjects who are pregnant or are planning to become pregnant during the study timeframe
3. previous ACL injury
4. previous surgery to either knee
5. bony fracture accompanying ACL injury
6. chronic ACL injuries (for our study, this is defined as patient reporting to a physician greater than 2 weeks after initial injury)
7. patients who experienced a knee dislocation
8. History of blood clots
9. Previous deep vein thrombosis
10. Use of estrogen or progestin contraceptive
11. History of cerebrovascular disease
12. History of peripheral vascular disease
13. History of Sickle Cell Anemia
14. History of chronic muscular disorder (e.g. fibromyalgia)
15. History of severe hypertension

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline to return to activity in quadriceps muscle strength | Pre-surgery (baseline), Return to Activity (~9 months post-surgery)
  concentric isokinetic muscle strength at 60 degrees per second

SECONDARY OUTCOMES:
Knee Flexion Angle | Return to Activity (~9 months post-surgery)
  Peak knee flexion angle recorded during a single-legged hop (units: degrees)
Knee Flexion Moment | Return to Activity (~9 months post-surgery)
  Peak knee flexion moment recorded during a single-legged hop (units: Nm/kg)
Change from baseline to pre-intervention in PROMIS Global Health Scale | Pre-surgery (baseline), Pre-intervention (~10 weeks post-surgery)
  Patient-reported outcome measured to assess health related quality of life. Physical Function Average: t score = 50±10 Min: 10 Max: 90
Change from baseline to post-intervention in PROMIS Global Health Scale | Pre-surgery (baseline), Post-intervention (~18 weeks post-surgery)
  Patient-reported outcome measured to assess health related quality of life. Physical Function Average: t score = 50±10 Min: 10 Max: 90
Change from baseline to return to activity in PROMIS Global Health Scale | Pre-surgery (baseline),Return to Activity (~9 months post-surgery)
  Patient-reported outcome measured to assess health related quality of life. Physical Function Average: t score = 50±10 Min: 10 Max: 90

OTHER OUTCOMES:
Change from baseline to pre-intervention in quadriceps cross-sectional area | Pre-surgery (baseline), Pre-intervention (~10 weeks post-surgery)
  cross-sectional area of the quadriceps muscle
Change from baseline to post-intervention in quadriceps cross-sectional area | Pre-surgery (baseline), Post-intervention (~18 weeks post-surgery)
  cross-sectional area of the quadriceps muscle
Change from baseline to return to activity in quadriceps cross-sectional area | Pre-surgery (baseline), Return to Activity (~9 months post-surgery)
  cross-sectional area of the quadriceps muscle

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curran MT, Bedi A, Mendias CL, Wojtys EM, Kujawa MV, Palmieri-Smith RM. Blood Flow Restriction Training Applied With High-Intensity Exercise Does Not Improve Quadriceps Muscle Function After Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Am J Sports Med. 2020 Mar;48(4):825-837. doi: 10.1177/0363546520904008. PMID 32167837